CLINICAL TRIAL: NCT00400621
Title: Assessment of Hepatic Injury in Subjects Who Consume Moderate Amounts of Alcohol While Being Administered Therapeutic Doses of Acetaminophen:
Brief Title: Effects of Therapeutic Doses of Acetaminophen in Moderate Drinkers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: COMIRB 02-999
Record Dates: First submitted 2006-11-16; First posted 2006-11-17 (Estimated); Last update posted 2024-07-08 (Actual); Status verified 2006-11

CONDITIONS: Moderate Alcohol Consumption (1-3 Drinks Per Day)
Keywords: acetaminophen; alcohol; liver injury
MeSH Terms: interventions — Acetaminophen

INTERVENTIONS:
Drug: acetaminophen

SUMMARY:
The study objective was to evaluate the safety of ten consecutive days of therapeutic acetaminophen dosing in moderate alcohol consumers. The main outcome was liver injury (measured by an increase in mean serum ALT or AST levels). Patients were randomly assigned to 10 days of acetaminophen or placebo. Blood tests were measured at baseline, day 4 and day 11 to look for injury. We hypothesized that there would be no difference in liver enzymes between the two groups.

ELIGIBILITY:
Inclusion criteria Adult volunteers of age 21 years or older, regardless of ethnicity or gender, who provided written consent and met all three of the following criteria of a moderate alcohol consumer:

1. Average baseline ethanol consumption of at least one alcoholic beverage per day before enrollment for the past two months. The estimate of ethanol intake was based on the average intake over seven days. For example, a person who ingested no alcohol on Sunday, Monday, Tuesday or Wednesday, two drinks on Thursday and four drinks on Friday and Saturday would be calculated as 10 drinks/7days = 1.4 drinks/day. The average alcoholic beverage contains 15 grams of alcohol(9).
2. Average baseline ethanol consumption of no more than three alcoholic beverages (> 45 grams of alcohol) per day, calculated as a weekly average over the preceding two months.
3. At least one alcohol-containing drink within the last 48 hours

Exclusion Criteria

Subjects were excluded from the study at baseline if any of the following were evident at baseline:

1. Serum acetaminophen level greater than 20 mcg/ml
2. Serum AST or ALT levels greater than 50 IU/L
3. If female, positive for b-HCG
4. Clinically intoxicated, psychiatrically impaired or unable to give informed consent
5. Known hypersensitivity to acetaminophen
6. History of ingesting more than four grams of acetaminophen per day for any of the four days preceding study enrollment
7. Alcoholic patients as defined by those who consume on average more than three alcoholic beverages daily
8. Currently enrolled in another trial or had been enrolled in another trial in the preceding three months

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2003-04; Study Completion 2003-09

PRIMARY OUTCOMES:
mean change in serum ALT between treatment groups

SECONDARY OUTCOMES:
proportion of patients that developed an abnormal ALT
proportion of patients that developed hepatoxicity (ALT>1000 IU>L)
proportion of patients that developed drug induced liver injury

CONTACTS AND LOCATIONS:
Overall Officials: Kennon Heard, MD, Principal Investigator — Rocky Mountain Poison Center